CLINICAL TRIAL: NCT02865798
Title: Multicenter Prospective Cohort Study of Senile Hospitalized Patients With Valvular Heart Disease
Brief Title: China Senile Valvular Heart Disease Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: VHD-20160805
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Heart Valve Diseases
Keywords: Heart Valve Diseases; Cardiovascular Diseases; Heart Disease; Valvular Heart Diseases
MeSH Terms: conditions — Heart Valve Diseases; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 6mL whole blood sample is collected in an EDTA vacuum tube.

SUMMARY:
Valvular heart diseases (VHD) are the most common causes of mortality and morbidity after coronary artery disease, hypertension, and heart failure, especially in senile patients who have more comorbidities and often require intervention. The prevalence of senile VHD is increased gradually as the growth of the age. In addition important changes have occurred as regards the presentation and treatment of the disease over recent years. However, there is little information about senile VHD in China. The purposes of this study are to evaluate the clinical characteristics, reasons for hospitalization, risk stratification, treatment modalities, quality of life and outcomes of senile hospitalized patients with VHD, to determine the risk factors affecting the prognosis, further to lay the foundation for establishing a prognosis model suitable for Chinese senile VHD.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients over 60 years old meet one of the following conditions.

* moderate or above valvular heart disease as defined by echocardiography:

  * aortic stenosis, moderate or above, or valve area ≤1.5cm2, or maximal jet velocity ≥3.0m/sec, or mean pressure gradient ≥20mmHg,
  * aortic regurgitation, moderate or above, or jet width ≥25% of left ventricular outflow tract, or regurgitant volume ≥30ml/beat, or regurgitant fraction ≥30%,
  * mitral stenosis, moderate or above, or valve area ≤2.0cm2,
  * mitral regurgitation, moderate or above, or effective regurgitant orifice ≥0.2cm2, or regurgitant volume ≥30ml/beat, or regurgitant fraction ≥30%,
  * tricuspid stenosis, moderate or above, or valve area ≤1.0cm2,
  * tricuspid regurgitation, moderate or above, or central jet area ≥5.0cm2,
  * pulmonic stenosis, moderate or above, or maximal jet velocity >4m/sec,
  * pulmonic regurgitation, moderate or above,
* or patients who had undergone any operation on a cardiac valve (percutaneous balloon commissurotomy, valve repair, valve replacement, transcatheter aortic valve implantation),
* or diagnosis of endocarditis as assessed by Duke criteria.

Exclusion Criteria:

* Patients cannot be followed up for any reasons.
* Patients in critical condition may be die in the near future.
* Patients have been enrolled in this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 71 hospitals have capable of valvular surgery in China, 4000 hospitalized patients over 60 years old with valvular heart disease will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao Q, Xu H, Liu Q, Ye Y, Zhang B, Li Z, Gao R, Wu Y. Therapeutic Decision-Making and Outcomes in Elderly Patients With Severe Symptomatic Aortic Stenosis: Prognostic Implications of Elderly Patients' Initial Decisions. Front Cardiovasc Med. 2021 Jul 26;8:696763. doi: 10.3389/fcvm.2021.696763. eCollection 2021. PMID 34381825